CLINICAL TRIAL: NCT00477451
Title: Investigation of a Single Dose of Staccato™ Alprazolam for Inhalation on Doxapram-Induced Panic Attack in Patients With Panic Disorder
Brief Title: Staccato Alprazolam in Panic Attack
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexza Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMDC-002-201
Record Dates: First submitted 2007-05-22; First posted 2007-05-23 (Estimated); Results first posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2008-06

CONDITIONS: Treatment of Induced Panic Attack
Keywords: Staccato™ Alprazolam, Panic Attack, Inhaled alprazolam
MeSH Terms: conditions — Panic Disorder | interventions — Doxapram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- RCT Placebo (Placebo Comparator): Subjects received inhaled placebo after 0.5 mg/kg doxapram IV in the randomized controlled trial
  Interventions: Drug: Inhaled placebo; Drug: IV doxapram
- RCT Alprazolam 1 mg (Experimental): Subjects received 1 mg inhaled Staccato alprazolam 10 s after 0.5 mg/kg doxapram IV in the randomized controlled trial
  Interventions: Drug: Inhaled alprazolam 1 mg; Drug: IV doxapram
- Open Label Inhaled Alprazolam 1 mg (Experimental): Subjects received 1 mg inhaled Staccato alprazolam 10 s after 0.5 mg/kg doxapram IV in the open label dose validation
  Interventions: Drug: Inhaled alprazolam 1 mg; Drug: IV doxapram
- Initial Inhaled Alprazolam 2 mg (Experimental): Subjects received 2 mg inhaled Staccato alprazolam 10 s after 0.5 mg/kg doxapram IV in the initial open label dose assessment
  Interventions: Drug: Inhaled alprazolam 2 mg; Drug: IV doxapram

INTERVENTIONS:
Drug: Inhaled placebo — Inhaled Staccato Alprazolam Placebo
  Arms: RCT Placebo
Drug: Inhaled alprazolam 1 mg — Inhaled Staccato Alprazolam 1 mg
  Arms: Open Label Inhaled Alprazolam 1 mg; RCT Alprazolam 1 mg
Drug: Inhaled alprazolam 2 mg — Inhaled Staccato Alprazolam 2 mg
  Arms: Initial Inhaled Alprazolam 2 mg
Drug: IV doxapram — 0.5 mg/kg doxapram IV approximately 10s after receiving inhaled alprazolam or placebo

SUMMARY:
We are developing Staccato™ Alprazolam for the treatment of Panic attacks associated with panic disorder. This study will provide an initial assessment of efficacy, and to continue to describe the tolerability and pharmacokinetics, of a single inhaled dose of Staccato Alprazolam on a doxapram-induced panic attack in patients with panic disorder.

DETAILED DESCRIPTION:
The study will be conducted at multiple centers. A total of 42 male and female panic disorder patients will be studied. The first 6 subjects will receive Staccato Alprazolam 1 mg open label to validate the dose selection. The remaining 36 subjects will be treated with either Staccato Alprazolam at the chosen dose; or with Staccato Placebo in a double blind, randomized order.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who meet DSM-IV criteria for panic disorder, with or without agoraphobia.
2. Subjects who have had at least one panic attack per week in each of the four weeks prior to the start of treatment and/or have a Mobility Inventory Score of 3.3 (alone) or 2.5 (accompanied).
3. Male or female subjects who are English-speaking between 18 and 55 years of age.
4. Female subjects who are not pregnant, or are surgically sterile or 2 years postmenopausal. If of childbearing potential, she must be using a medically-accepted method of birth control and agree to continue use of this method for at least 30 days after the study (i.e., barrier method with spermicide, steroidal contraceptive [oral, transdermal, and implanted, including Depo-Provera; contraceptives must be used in conjunction with a barrier method], or intrauterine device).
5. Subjects who are medically healthy (i.e. without a clinically significant unstable medical condition such as asthma, coronary artery disease, renal insufficiency, etc.)
6. Subjects who are able to give informed consent for participation.
7. Subjects who are able to be withdrawn from current panic disorder medication because it is ineffective.

Exclusion Criteria:

1. Subjects who have met DSM-IV criteria for substance abuse or dependence within six months of study entry must be excluded.
2. Subjects with a baseline Acute Panic Inventory (22 item test) score of 41 or higher on the test day must be excluded.
3. Subjects who are taking benzodiazepines, SSRIs, or medication that is effective for the prevention or treatment of the patient's panic disorder (i.e., no patient will be withdrawn for medication that is working for the purpose of entry into this study) must be excluded.
4. Subjects who are clinically depressed must be excluded.
5. Subjects who have received an investigational drug within 30 days (or within 5 half lives of the investigational drug) prior to test day must be excluded.
6. Subjects with epilepsy or other convulsive disorders must be excluded.
7. Subjects with a history of allergy or intolerance to benzodiazepines or related drugs (alprazolam, lorazepam, diazepam, etizolam, clonazepam, adinazolam) must be excluded.
8. Subjects who test positive for alcohol or have a positive urine drug screen for illicit or disallowed drugs must be excluded. Subjects should refrain from consuming alcohol for at least 48 hours prior to dosing.
9. Female subjects who are breastfeeding or have a positive pregnancy test must be excluded.
10. Subjects who have any other disease or condition, by history, physical examination, or laboratory abnormalities that in the investigator's opinion, would present undue risk to the subject, or may confound the interpretation of study results must be excluded.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2007-05 (Actual); Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Mathew, MD, Principal Investigator — Mt. Sinai School of Medicine; Jeremy Coplan, MD, Principal Investigator — State University of New York - Downstate Medical Center; Laszlo Papp, MD, Principal Investigator — New York State Psychiatric Institute
Locations (3):
- United States (3):
  - SUNY Downstate Medical Center, Brooklyn, New York
  - New York State Psychiatric Institute, New York, New York
  - Mt. Sinai School Of Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
IPD submitted to regulatory authorities. Others may contact Alexza Pharmaceuticals, Inc. Please send your request to ClinicalTrialsInfo@alexza.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RCT Placebo | RCT Alprazolam 1 mg | Open Label Inhaled Alprazolam 1 mg | Initial Inhaled Alprazolam 2 mg
Started | 20 | 20 | 7 | 2
Completed | 20 | 20 | 7 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | RCT Placebo | RCT Alprazolam 1 mg | Open Label Inhaled Alprazolam 1 mg | Initial Inhaled Alprazolam 2 mg | Total
Number analyzed (Participants) | 20 | 20 | 7 | 2 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 7 | 2 | 49
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (10.2) | 32.1 (9.45) | 43.1 (13.6) | 37.5 (0.707) | 34.3 (10.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 1 | 1 | 23
  Male | 11 | 8 | 6 | 1 | 26
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 7 | 2 | 49

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Doxapram-induced Panic Attack
Description: doxapram-induced panic attack of sufficient intensity (DIPASI) defined as a 10 or greater increase from baseline in the acute panic inventory (API)
Time Frame: 0 to 2 hours
Population: RCT Population (N=40)
Measure: Count of Participants; unit: Participants
Arm/Group | RCT Placebo | RCT Alprazolam 1 mg
Number analyzed (Participants) | 20 | 20
Participants | 14 | 9
Statistical Analysis 1: Comparison: RCT Placebo vs RCT Alprazolam 1 mg; Test type: Superiority; p = 0.200, Fisher Exact

2. Primary Outcome: Duration of the Doxapram-induced Panic Attack
Description: Length of time from the doxapram injection to the time at which the acute panic inventory (API) value returns to within 10 points of the baseline API value. 0=never exceeded 0, 61=exceeded by more than 10 points still at end of assessment of 60 minutes. Thus each would have a duration whether or not they had a panic attack (DIPASI)
Time Frame: 1 hr post-dose
Population: RCT Population (N=40)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | RCT Placebo | RCT Alprazolam 1 mg
Number analyzed (Participants) | 20 | 20
minutes | 12.2 (17.2) | 9.25 (14.1)
Statistical Analysis 1: Comparison: RCT Placebo vs RCT Alprazolam 1 mg; Test type: Superiority; p = 0.368, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Borg Max Change From Baseline
Description: Subjects asked to "Point to the number (0 to 10) which matches how breathless you feel now" where 0=nothing at all to 10=very, very strong
Time Frame: 45 minutes
Population: RCT Population (N=40)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RCT Placebo | RCT Alprazolam 1 mg
Number analyzed (Participants) | 20 | 20
units on a scale | 5.73 (2.85) | 4.63 (2.56)
Statistical Analysis 1: Comparison: RCT Placebo vs RCT Alprazolam 1 mg; Test type: Superiority; p = 0.207, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were considered treatment related from the first exposure to study treatment until 30 days after the last treatment
Description: Adverse events (AEs) were assessed predose and at 13 pre-specified time points as well as whenever spontaneously reported by the subjects or study staff
Arm/Group | RCT Placebo | RCT Alprazolam 1 mg | Open Label Inhaled Alprazolam 1 mg | Initial Inhaled Alprazolam 2 mg
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/7 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/7 | 0/2
Other Adverse Events (participants affected / at risk) | 2/20 | 11/20 | 1/7 | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RCT Placebo (N=20) | RCT Alprazolam 1 mg (N=20) | Open Label Inhaled Alprazolam 1 mg (N=7) | Initial Inhaled Alprazolam 2 mg (N=2)
Dysgeusia (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SEDATION (Nervous system disorders) | 2 (2) | 9 (9) | 1 (1) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less